CLINICAL TRIAL: NCT04916834
Title: Impact of SARS-CoV-2/COVID-19 Related Pneumonia on Lung Function and Structure - Prospective Case Control Study
Brief Title: Impact of Severe Acute Respiratory Syndrome (SARS-CoV-2/COVID-19) Related Pneumonia on Lung Function and Structure.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute for Tuberculosis and Lung Diseases, Poland (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: IGICHP/7.52
Record Dates: First submitted 2020-11-09; First posted 2021-06-08 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Covid19; SARS-CoV Infection; Pulmonary Function; Pneumonia, Viral
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective study in a group of patients with COVID-19 pneumonia.

DETAILED DESCRIPTION:
Objective:

Assessment of pulmonary and heart dysfunction, fibrosis-related markers and antibodies as well as the search for risk factors for an unfavorable course and possible complications in patients after pneumonia due to SARS-CoV-2 (COVID-19) infection.

Patients:

A group of approx. 100 patients assessed shortly after pneumonia and followed up, investigated after 3 and 6 months with possible prolongation to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed SARS-CoV-2 infection with pneumonia hospitalized
2. Two negative PCR results of a swab from the respiratory tract in succession, including the last one taken no later than 3 days before the planned lung function tests (1st visit).

Exclusion Criteria:

1. Lack of patient consent,
2. Present contraindications for lung function tests
3. Inability to perform correctly lung function measurements

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients dicharged after confirmed COVID-19 pneumonia (positive PCR and lung involvement in HRCT, hospitalized)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in lung transfer factor for carbon monoxide (TL,CO) at 3, 6 and 12 months after COVID-19 pneumonia | 0, 3, 6, 12 months after COVID-19 pneumonia
  Lung transfer factor for carbon monoxide (TL,CO) will be measured using single breath method, results will be reported as absolute values (mmol/min/kPa)
Change from baseline in lung transfer factor for carbon monoxide (TL,CO) at 3, 6 and 12 months after COVID-19 pneumonia | 0, 3, 6, 12 months after COVID-19 pneumonia
  Lung transfer factor for carbon monoxide (TL,CO) will be measured using single breath method, results will be reported as % of predicted using GLI-2017 references
Change from baseline in forced vital capacity (FVC) at 3, 6 and 12 months after COVID-19 pneumonia | 0, 3, 6, 12 months after COVID-19 pneumonia
  Forced vital capacity (FVC) will be measured using spirometry according to ATS/ERS 2019 guidelines, results will be reported as absolute values (L)
Change from baseline in forced vital capacity (FVC) at 3, 6 and 12 months after COVID-19 pneumonia | 0, 3, 6, 12 months after COVID-19 pneumonia
  Forced vital capacity (FVC) will be measured using spirometry according to ATS/ERS 2019 guidelines, results will be reported as % of predicted using GLI-2012 references
Change from baseline in forced expiratory volume at 1 second (FEV1) at 3, 6 and 12 months after COVID-19 pneumonia | 0, 3, 6, 12 months after COVID-19 pneumonia
  Forced expiratory volume at 1 second (FEV1) will be measured using spirometry according to ATS/ERS 2019 guidelines, results will be reported as absolute values (L)
Change from baseline in forced expiratory volume at 1 second (FEV1) at 3, 6 and 12 months after COVID-19 pneumonia | 0, 3, 6, 12 months after COVID-19 pneumonia
  Forced expiratory volume at 1 second (FEV1) will be measured using spirometry according to ATS/ERS 2019 guidelines, results will be reported as % of predicted using GLI-2012 references
Change from baseline in total lun capacity (TLC) at 3, 6 and 12 months after COVID-19 pneumonia | 0, 3, 6, 12 months after COVID-19 pneumonia
  Total lung capacity will be measured using body plethysmography method according to ATS/ERS 2005 guidelines, results will be reported as absolute values (L)
Change from baseline in total lun capacity (TLC) at 3, 6 and 12 months after COVID-19 pneumonia | 0, 3, 6, 12 months after COVID-19 pneumonia
  Total lung capacity will be measured using body plethysmography method according to ATS/ERS 2005 guidelines, results will be reported as % of predicted using most recent references
Change in prevalence of abnormal (low) lung transfer factor for carbon monoxide (TL,CO) results at 3, 6 and 12 months after COVID-19 pneumonia | 0, 3, 6, 12 months after COVID-19 pneumonia
  Abnormal (low) lung transfer factor for carbon monoxide (TL,CO) will be identified with cut-off point at the level of 5th percentile (-1.64 SD) using most recent predicted values (GLI-2017), prevalence will be reported as % of investigated group
Change in prevalence of obstructive ventilatory impairment at 3, 6 and 12 months after COVID-19 pneumonia | 0, 3, 6, 12 months after COVID-19 pneumonia
  Obstructive ventilatory impairment (airway obstruction) will be identified with FEV1/FVC ratio below lower limit of normal, cut-off point at the level of 5th percentile (-1.64 SD) will be used with most recent predicted values (GLI-2012), prevalence will be reported as % of investigated group
Change in prevalence of restrictive ventilatory impairment at 3, 6 and 12 months after COVID-19 pneumonia | 0, 3, 6, 12 months after COVID-19 pneumonia
  Restrictive ventilatory impairment will be identified with total lung capacity (TLC) below lower limit of normal, cut-off point at the level of 5th percentile (-1.64 SD) will be used with most recent predicted values, prevalence will be reported as % of investigated group
Change in lung structure from the baseline | 3, 6, 12 months
  Change in lung structure will be assessed using high resolution computed tomography (HRCT) performed at 3, 6 and 12 months after initial investigation. Quantitive assessment of abnormalities will be performed and compared with initial investigation performed during acute phase of COVID-19 pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr W Boros, MD, PhD, Principal Investigator — National TB & Lung Diseases Research Institute
Locations (1):
- National Institute for Tuberculosis and Lung Diseases, Warsaw, Masovian Voivodeship, Poland